CLINICAL TRIAL: NCT01457573
Title: Urinary Nerve Growth Factor as a Biomarker for Medical Treatment of Male Lower Urinary Tract Symptoms: A Pilot Trial
Brief Title: Pilot Trial Of Urinary Nerve Growth Factor (NGF) As Biomarker for Male Lower Urinary Tract Symptoms
Acronym: LUTS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Timothy Boone, MD, PhD (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Timothy Boone, MD, PhD, Sponsor-Investigator/Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00006253; IRB# 0711-0124 (Other: HMRI IRB)
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Tamsulosin; Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- One (single arm) (Experimental): All men will receive morning dosing with Tamsulosin (Flomax) 0.4 mg (1 tab) and Solifenacin (Vesicare) 5 mg (1 tab) orally at the same time.
  Interventions: Drug: Tamsulosin; Drug: Solifenacin

INTERVENTIONS:
Drug: Tamsulosin — Alpha blocker used to in the treatment of urinary difficulties related to enlarged prostate or symptomatic benign prostatic hypertrophy. All men will receive Tamsulosin (Flomax®) 0.4 mg, 1 tab, per morning with Solifenacin (Vesicare®).
  Other Names: tamsulosin hydrochloride, tamsulosin HCl, Flomax®
Drug: Solifenacin — Antispasmodic/anticholinergic used to treat overactive bladder. All men will receive Solifenacin (Vesicare®) 5 mg, 1 tab, per morning with Tamsulosin.
  Other Names: solifenacin succinate, VESIcare®, Vesicare®

SUMMARY:
A single center, pilot trial using tamsulosin and solifenacin in 10 men with symptomatic lower urinary tract symptoms (LUTS). Subjects will be evaluated at baseline, 1, 2, and 3 months for urinary NGF, urine creatinine, NGF/CR ratio and patient reported outcomes through questionnaires.

DETAILED DESCRIPTION:
Single center, pilot trial, single arm study using once daily dosing of tamsulosin and solifenacin in 10 men with symptomatic lower urinary tract symptoms (LUTS). Assessments occur at Baseline, 1 Month, 2 Month and 3 Month to evaluate: urinary NGF (pg/mL), urine creatinine (mg/dL), NGF/Cr ratio and patient reported questionnaire outcomes (AUA Symptom Score/IPSS, Patient Perception of Bladder Condition, Patient Perception of Urge Intensity 'PPIUS', LUTS Urinary Symptoms and Quality of Life). Each participant is assessed from baseline to Month 3 measurements. Protection of human subjects will be provided through the Houston Methodist Research Institute Institutional Review Board (see appendix 2). All men will receive morning dosing with Tamsulosin 0.4 mg (1 tab) and Solifenacin 5 mg (1 tab) orally at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Men > 45 years old with symptomatic LUTS (clinical benign prostatic hypertrophy/BPH)
* International Prostate Symptom Score (IPSS) > 8
* PSA < 10 ng/ml (negative biopsies within 6 months for any age-specific PSA elevation suspicious for prostate carcinoma)
* Post void residual urine < 150 mls
* Urinary Flow rate > 15 mL/sec

Exclusion Criteria:

* Neurogenic bladder
* Urinary tract infection, Urinary stone(s), Urinary tract tumor
* Radiation therapy for urologic malignancy or prostate surgery; radiation to pelvic, colon, rectum, prostate, bladder, uterus or ovaries
* Alpha blocker therapy or anticholinergic therapy within 3 months of entry or 5 alpha reductase therapy within 18 months.
* History of cataracts with planned surgery

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Boone, MD,PhD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- The Methodist Hospital System, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Plan to share data to be determined.

REFERENCES:
- [Background] McVary KT. 2010 AUA Benign Prostatic Hyperplasia Clinical Guidelines. Panel Chair, AUA News 2010; 15 (3) 10 - 11.
- [Background] Chapple CR, Roehrborn CG. A shifted paradigm for the further understanding, evaluation, and treatment of lower urinary tract symptoms in men: focus on the bladder. Eur Urol. 2006 Apr;49(4):651-8. doi: 10.1016/j.eururo.2006.02.018. Epub 2006 Feb 17. PMID 16530611
- [Background] Kaplan SA. New data on Tolterodine: Do recent findings dispel questions about treating overactive bladder in men? Eur Urology 2007; Suppl 6: 10-16.
- [Background] Lee JY, Kim HW, Lee SJ, Koh JS, Suh HJ, Chancellor MB. Comparison of doxazosin with or without tolterodine in men with symptomatic bladder outlet obstruction and an overactive bladder. BJU Int. 2004 Oct;94(6):817-20. doi: 10.1111/j.1464-410X.2004.05039.x. PMID 15476515
- [Background] Kaplan SA, Roehrborn CG, Rovner ES, Carlsson M, Bavendam T, Guan Z. Tolterodine and tamsulosin for treatment of men with lower urinary tract symptoms and overactive bladder: a randomized controlled trial. JAMA. 2006 Nov 15;296(19):2319-28. doi: 10.1001/jama.296.19.2319. PMID 17105794
- [Background] Kaplan SA, Roehrborn CG, Chancellor M, Carlsson M, Bavendam T, Guan Z. Extended-release tolterodine with or without tamsulosin in men with lower urinary tract symptoms and overactive bladder: effects on urinary symptoms assessed by the International Prostate Symptom Score. BJU Int. 2008 Nov;102(9):1133-9. doi: 10.1111/j.1464-410X.2008.07761.x. Epub 2008 May 26. PMID 18510659
- [Background] Kaplan SA, Goldfischer ER, Steers WD, Gittelman M, Andoh M, Forero-Schwanhaeuser S. Solifenacin treatment in men with overactive bladder: effects on symptoms and patient-reported outcomes. Aging Male. 2010 Jun;13(2):100-7. doi: 10.3109/13685530903440408. PMID 20001469
- [Background] Liu HT, Kuo HC. Urinary nerve growth factor level could be a potential biomarker for diagnosis of overactive bladder. J Urol. 2008 Jun;179(6):2270-4. doi: 10.1016/j.juro.2008.01.146. Epub 2008 Apr 18. PMID 18423678
- [Background] Yokoyama T, Kumon H, Nagai A. Correlation of urinary nerve growth factor level with pathogenesis of overactive bladder. Neurourol Urodyn. 2008;27(5):417-20. doi: 10.1002/nau.20519. PMID 17924444
- [Background] Liu HT, Chancellor MB, Kuo HC. Decrease of urinary nerve growth factor levels after antimuscarinic therapy in patients with overactive bladder. BJU Int. 2009 Jun;103(12):1668-72. doi: 10.1111/j.1464-410X.2009.08380.x. Epub 2009 Feb 11. PMID 19220267
- [Background] Jacobs BL, Smaldone MC, Tyagi V, Philips BJ, Jackman SV, Leng WW, Tyagi P. Increased nerve growth factor in neurogenic overactive bladder and interstitial cystitis patients. Can J Urol. 2010 Feb;17(1):4989-94. PMID 20156378
- [Background] Cardozo L, Hessdorfer E, Milani R, Arano P, Dewilde L, Slack M, Drogendijk T, Wright M, Bolodeoku J; SUNRISE Study Group. Solifenacin in the treatment of urgency and other symptoms of overactive bladder: results from a randomized, double-blind, placebo-controlled, rising-dose trial. BJU Int. 2008 Nov;102(9):1120-7. doi: 10.1111/j.1464-410X.2008.07939.x. Epub 2008 Oct 6. PMID 18990175
- [Result] Dmochowski RR, Gomelsky A. Overactive bladder in males. Ther Adv Urol. 2009 Oct;1(4):209-21. doi: 10.1177/1756287209350383. PMID 21789068

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were approached by the PI and Study Team in an outpatient urology clinic setting between October 2011 and December 2014 for recruitment to the male lower urinary tract symptoms study.
Groups:
- Single Arm (Tamsulosin and Solifenacin): 10 Men with lower urinary tract symptoms (LUTS), consistent with BPH, were screened in our urology clinics for participation in a clinical trial.
Period: Overall Study
Arm/Group | Single Arm (Tamsulosin and Solifenacin)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Men > 50 years old with urinary frequency symptoms, who entered study not taking any bladder related medications and on study took tamsulosin and solifenacin orally everyday throughout the study with follow-up assessments at Month 1/week 4, Month 2 week 8, and Month 3/week 12.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] | 64 [48 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 10
Baseline Post-void residual (PVR) of urine [Mean (Standard Deviation); unit: ml] — PVR is the measure of urine measured in milliliters (ml), by an ultrasound over the abdomen, to measure how much urine remains in the bladder after it is completely empty following urodynamic measurements. Urodynamics is the test done right before the PVR to measure how fast and how much, volume of urine is emptied from the bladder. These measurements help identify issues related to enlarged prostate or other issue.
  ml | 53.89 (51.74)
Baseline Maximum urinary flow rate [Mean (Standard Deviation); unit: ml/s] — Max urinary flow rate in ml/sec measured by urodynamics at baseline. An average rate in males is 21 ml/sec (ages 14-45 years-old) and 12 ml/sec in males (ages 46-65 years-old).
  ml/s | 18.71 (9.27)
Baseline International Prostate Symptom Score (IPSS) [Mean (Standard Deviation); unit: units on a scale] — IPSS is a questionnaire, max of 35 points, none (0), to few symptoms to 35 (symptomatic), administered at baseline, which measures incomplete bladder emptying, frequency, urgency, straining, and nocturia.
  units on a scale | 18.2 (5.07)
Baseline Patient Perception of Urgency Score (PPUS) [Mean (Standard Deviation); unit: units on a scale] — PPUS is in questionnaire format with a max score of 4. Subject have a single rating, low score (none) to 4 (symptoms).
  units on a scale | 2.5 (0.85)
Baseline Perception of Bladder Condition (PBC) [Mean (Standard Deviation); unit: units on a scale] — Perception of bladder control measured in questionnaire format with single max rating up to 6, comparing baseline. Low score (none) to 6 (symptoms).
  units on a scale | 3.5 (0.85)
Baseline International Consultation on Incontinence Mod. Questions-Male Lower Urinary Tract Symptoms [Mean (Standard Deviation); unit: units on a scale] — ICIQ MLUTS (max score = 182) quality of life questionnaire to measure baseline. Low score (none to few symptoms) to 182 (very symptomatic).
  units on a scale | 67.2 (21.04)
Baseline International Consultation on Incontinence Mod. Questions Lower Urinary Tract Symptoms QoL [Mean (Standard Deviation); unit: units on a scale] — ICIQ LUTs Quality of Life with max score = 288 from a questionnaire taken at baseline. Low score (none to few symptoms) to 288 (very symptomatic).
  units on a scale | 122.6 (59.53)
Baseline Urinary Nerve Growth Factor (pg/ml)/Cr (mg/dl) [Mean (Standard Deviation); unit: ratio] — Urinary Nerve Growth Factor (uNGF) from a biomarker in pg/ml in a ratio over urinary creatinine (u-Cr) obtained from a lab tested urinalysis in mg/dl.
  ratio | 34.20 (56.69)
Baseline Urinary Nerve Growth Factor [Mean (Standard Deviation); unit: pg/ml] — Urine collected for urinary nerve growth factor (u-NGF with units: pg/ml) measurement at baseline.
  pg/ml | 37.10 (21.24)

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary Nerve Growth Factor (pg/mL) at Baseline Compared to Post Dose Exposure at Mo.3/Wk12
Description: Urine sample tested for urinary Nerve Growth Factor (uNGF as measured in pg/mL), a small secreted protein in the bladder that supports bladder function regulation, at baseline (pre-dose) and week 12/Month 3 post-dose, after using daily tamsulosin and solifenacin.
Time Frame: Change from baseline to week 12 (3 months)
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Single Arm Receiving Tamsulosin 0.4 mg and Solifenacin 5 mg: All men will receive morning dosing with Tamsulosin (Flomax) 0.4 mg and Solifenacin (Vesicare) 5 mg orally at the same time.
  Solifenacin (Vesicare) 5 mg orally at the same time.: Drug: Tamsulosin 0.4 mg in combination with Solifenacin 5 mg
  All men will receive morning dosing with Tamsulosin (Flomax) 0.4 mg and Solifenacin (Vesicare) 5 mg orally at the same time.
Arm/Group | Single Arm Receiving Tamsulosin 0.4 mg and Solifenacin 5 mg
Number analyzed (Participants) | 10
pg/ml | -10.9 (22.81)

2. Primary Outcome: Change From Baseline in Urinary Growth Factor to Creatinine Ratio (GF/Cr)
Description: The urinary growth factor (GF) to creatinine ratio may be potential biomarker for overactive bladder, based on published articles. Measuring the ratio at baseline and Month 3, comparing the difference after treatment with tamsulosin and solifenacin which may provide insight into how lower urinary tract symptoms in men progresses.
Time Frame: change from baseline score to Month 3
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Baseline Characteristics: Men > 50 years old with symptomatic LUTS (IPSS > 8), PSA < 10, PVR < 150 mls and maximum urinary flow rate > 10 mls/sec could enter the trial.
Arm/Group | Baseline Characteristics
Number analyzed (Participants) | 10
ratio | -19.61 (13.21)

3. Secondary Outcome: Change in Post Void Residual (mL) at Baseline Compared to Post Dose Exposure at Mo.1, Mo, 2, and Mo. 3/Wk12
Description: Urine sample tested for urinary post void residual (measured in mL) at baseline (pre-dose), Month 1 and Month 2and week 12/Month 3 post-dose, post dose w/tamsulosin and solifenacin.
Time Frame: Change from baseline to months 1, 2 and 3
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Single Arm Receiving Tamsulosin 0.4 mg and Solifenacin 5 mg
Number analyzed (Participants) | 10
ml
  Change at Month 1 | -6.90 (90.58)
  Change at Month 2 | -10.00 (60.84)
  Change at Month 3 | -3.60 (92.71)

4. Secondary Outcome: Change in Maximum Urinary Flow Rate (ml/s) at Baseline Compared to Post Dose Exposure at Mo.1, Mo, 2, and Mo. 3/Wk12
Description: Urination flow rate (measured in milliliters per second) at baseline (pre-dose), and Month 1, Month 2, and Month 3/Week 12 pose-dosing with tamsulosin and solifenacin. An average maximum urinary flow rate in males is 21 ml/sec aged 14-45 years-old and 12 ml/sec in males aged 46-65 years-old.
Time Frame: Change from baseline to months 1, 2 and 3
Measure: Mean (Standard Deviation); unit: ml/s
Arm/Group | Single Arm Receiving Tamsulosin 0.4 mg and Solifenacin 5 mg
Number analyzed (Participants) | 10
ml/s
  Change at Month 1 | -3.20 (6.37)
  Change at Month 2 | -3.90 (9.16)
  Change at Month 3 | -4.70 (9.38)

5. Secondary Outcome: Change in IPSS-International Prostate Score Scale at Baseline Compared to Post Dose Survey at Month 1, 2, and Month 3/Week12.
Description: The survey, IPSS-International Prostate Score Scale, survey responses measured 0-35, is collected at baseline compared to post dose survey response at Month 1, Month 2, and Month 3/Week12 post-dose. The lower the score is indicative of less or fewer urinary symptoms while 35 is consistent with more bothersome symptoms.
Time Frame: Change from baseline to months 1, 2 and 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm Receiving Tamsulosin 0.4 mg and Solifenacin 5 mg
Number analyzed (Participants) | 10
units on a scale
  Change at Month 1 | -2.00 (8.82)
  Change at Month 2 | -5.30 (6.40)
  Change at Month 3 | -7.33 (6.98)

6. Secondary Outcome: Change in PPUS-Patient Perception of Urinary Urgency Survey Score at Baseline Compared to Post Dose Exposure at Mo.1, Mo, 2, and Mo. 3/Wk12
Description: The Patient Perception of Urinary Urgency self administered survey score has a maximum score 4, zero to four, for how severe a patient describes their urinary voiding frequency. Four is the most bothersome score, 0 or 1 is the least bothersome. Pre-dose / baseline score is compared at Month 1, Month 2, and Month 3, after dosing with tamsulosin and solifenacin.
Time Frame: Change from baseline to months 1, 2 and 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm Receiving Tamsulosin 0.4 mg and Solifenacin 5 mg
Number analyzed (Participants) | 10
units on a scale
  Change at Month 1 | 0.00 (0.67)
  Change at Month 2 | 0.30 (0.67)
  Change at Month 3 | 0 (1.41)

7. Secondary Outcome: Change in PBC-Patient Perception of Bladder Condition at Baseline Compared to Post Dose Exposure at Mo.1, Mo, 2, and Mo. 3/Wk12
Description: Change in the Perception of Bladder through a self administered survey at baseline compared to Month 1, Month 2, and Month 3, following exposure to tamsulosin and solifenacin. The survey score measures from zero to 6, with 6 being the most bothersome bladder symptoms and 0 to 1 being the least bothersome.
Time Frame: Change from baseline to months 1, 2 and 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm Receiving Tamsulosin 0.4 mg and Solifenacin 5 mg
Number analyzed (Participants) | 10
units on a scale
  Change at Month 1 | 1.29 (1.25)
  Change at Month 2 | 0.29 (1.11)
  Change at Month 3 | 0.00 (0.82)

8. Secondary Outcome: Change in ICIQ-MLUTS - International Consultation on Incontinence Modular Questionnaire for Male LUTS Baseline Compared to Post Dose Exposure at Mo.1, Mo, 2, and Mo. 3/Wk12
Description: Measuring change in the International Consultation on Incontinence Modular Questionnaire for male lower urinary tract symptoms through a self administered survey at baseline compared to Month 1, Month 2, and Month 3, after exposure to tamsulosin and solifenacin. The survey score is a zero to 182 range with 182 being the most bothersome and zero to one being the least bothersome.
Time Frame: Change from baseline to months 1, 2 and 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm Receiving Tamsulosin 0.4 mg and Solifenacin 5 mg
Number analyzed (Participants) | 10
units on a scale
  Change at Month 1 | -22.40 (16.98)
  Change at Month 2 | -22.20 (16.88)
  Change at Month 3 | -29.8 (25.97)

9. Secondary Outcome: Change in ICIQ LUTS QoL -International Consultation on Incontinence Modular Questionnaire LUTS Quality of Life for Male LUTS Baseline Compared to Post Dose Exposure at Mo.1, Mo, 2, and Mo. 3/Wk12
Description: Change in the International Consultation on Incontinence Modular Questionnaire on lower urinary tract symptoms quality of life survey for men, self administered, compared to Month 1, Month 2, and Month 3, after exposure to tamsulosin and solifenacin. The survey scoring is zero to 182, with 182 being the most bothersome and 0 to 1 being the least bothersome.
Time Frame: Change from baseline to months 1, 2 and 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm Receiving Tamsulosin 0.4 mg and Solifenacin 5 mg
Number analyzed (Participants) | 10
units on a scale
  Change at Month 1 | 34.60 (37.61)
  Change at Month 2 | 38.30 (33.15)
  Change at Month 3 | -9.00 (37.59)

10. Secondary Outcome: Change in Urinary Nerve Growth Factor (pg/mL) at Baseline Compared to Post Dose Exposure at Mo.1/Wk4 and Mo.2/Wk8
Description: Urine sample tested for urinary Nerve Growth Factor (uNGF as measured in pg/mL), a small secreted protein in the bladder that supports bladder function regulation, at baseline (pre-dose) compared to Month 1/Week 4 and Month 2/Week 8, post dosing with tamsulosin and solifenacin.
Time Frame: Change from baseline to Mo.1/Wk4 and Mo.2/Wk8
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Single Arm Receiving Tamsulosin 0.4 mg and Solifenacin 5 mg
Number analyzed (Participants) | 10
pg/ml
  Change at Month 1 | 11.17 (22.68)
  Change at Month 2 | 15.64 (38.76)

11. Secondary Outcome: Change in Urinary Growth Factor to Creatinine Ratio (GF/Cr) From Baseline Compared to Month 1/Week4 and Month 2/Week 8.
Description: Assessing the change from baseline to Month 1/Week 4 and Month 2/Week 8, of the urinary growth factor (GF) to creatinine ratio in men, which may be potential biomarker for overactive bladder, based on published articles. Measuring the ratio at baseline compared to Month 1 and Month 2 may provide insight into how lower urinary tract symptoms in men progresses.
Time Frame: change from baseline score to Mo.1/Wk4 and Mo.2/Wk8 scores
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Baseline Characteristics
Number analyzed (Participants) | 10
ratio
  Change at Month 1 | -21.85 (14.23)
  Change at Month 2 | -20.56 (18.96)

ADVERSE EVENTS:
Time Frame: 3 years
Description: All reported events were assessed by the Principal Investigator and resulted in no withdrawals due to study medications.
Groups:
- Participant Flow: 10 Men with lower urinary tract symptoms (LUTS), consistent with BPH, were screened in our urology clinics for participation in a clinical trial.
Arm/Group | Participant Flow
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participant Flow (N=10)
Fatigue (General disorders) | 1 (1) — Mild fatigue requiring no treatment (S#02)
malaise (General disorders) | 1 (1) — Mild malaise requiring no treatment (S#02).
bloating (Gastrointestinal disorders) | 1 (1) — Mild bloating lasting two weeks and not requiring treatment (S#02).
blurred vision (Eye disorders) | 1 (1) — Mild blurred vision not requiring treatment or intervention (S#02).
decreased memory (Nervous system disorders) | 1 (1) — Mild memory decrease, not requiring treatment or intervention (S#06).
urinary frequency (Renal and urinary disorders) | 1 (1) — Mild increase in urinary frequency not requiring medication or treatment which resolved after six weeks (S#06).
constipation (Gastrointestinal disorders) | 1 (2) — Moderate constipation, resolved with over-the-counter stool softener, 3 months duration (S#07) and Mild constipation resolving after 2 weeks without treatment (S#10).
tinnitus (Ear and labyrinth disorders) | 1 (1) — Mild ringing in ears, resolved after 14 days without treatment or intervention (S#07).
reduced ejaculation (Reproductive system and breast disorders) | 1 (1) — Reduced ejaculation (subjective report of moderate) but requiring no treatment or intervention while on study (S#07).
indigestion (Gastrointestinal disorders) | 1 (1) — Moderately increased indigestion (baseline/pre-study condition) treated with over-the-counter antacids while on study (S#09).
dry mouth (Skin and subcutaneous tissue disorders) | 1 (1) — Mild dry mouth lasting three weeks requiring no treatment or intervention (S#10).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less